CLINICAL TRIAL: NCT05781646
Title: Xpert MTB/RIF Assay for Diagnosis of Tuberculous Meningitis (TBM) in Maharaj Nakorn Chiang Mai Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Poramed Winichakoon, Physician, Chiang Mai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CMUXpertTBM
Record Dates: First submitted 2017-03-29; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Tuberculous Meningitis
Keywords: Xpert MTB/RIF; Tuberculous Meningitis
MeSH Terms: conditions — Tuberculosis, Meningeal

STUDY DESIGN:
Intervention Model Description: All patients older than 15 years old with subacute lymphocytic meningitis presenting to the internal medicine clinics of Maharaj Nakorn Chiang Mai hospital between January 2015 and March 2016 were recruited for the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Xpert (Experimental): Centrifuged CSF sent for Xpert MTB/RIF
  Interventions: Diagnostic Test: Xpert MTB/RIF

INTERVENTIONS:
Diagnostic Test: Xpert MTB/RIF — CSF samples was centrifuged at 3,000 - 4,000 X g for 15 minutes. Supernatant was removed to leave a 1-ml precipitate, which was then used for Ziehl-Neelsen AFB staining (100 μl), inoculation of MGIT culture (100 μl), and Xpert MTB/RIF testing (800 μl).

SUMMARY:
Early diagnosis and appropriate treatment of tuberculous meningitis (TBM) are crucial steps to reduce morbidity and mortality. The WHO recommended to use Xpert MTB/RIF assay to diagnose pulmonary TB, pediatrics TB, extra pulmonary TB and rifampicin resistance. However, the data of accuracy in diagnosis of TBM is still lacking. This study aimed to find out the diagnostic performance of Xpert MTB/RIF assay for the diagnosis of tuberculous meningitis, especially in patients who presented with subacute lymphocytic meningitis.

DETAILED DESCRIPTION:
Tuberculous meningitis (TBM) was the most serious manifestation of Mycobacterium tuberculosis infection with high rates of morbidity and mortality if treatment is delayed, especially in HIV-infected patients. The fatality rates increased to 60 percent compared to about one third in non-HIV infection. Prevalence and incidence of TBM worldwide is unclear. In 2015, the incidences of TBM were approximately 6-10 percent. In Northern Thailand, from the national survey programs, the prevalence rates of TBM were about 9.7 per 100,000 people, and TBM was the most common cause of death in extra-pulmonary TB patients with mortality rates about 0.54 per 100,000 people. However, these may be underreported due to diagnostic problems.

Prompt and accurate diagnoses with early treatments, were the key elements to reduce deaths and disabilities in TBM. However, there were some major obstacles in the diagnostic procedures concerning the limitations, such as low sensitivity in conventional acid-fast bacilli (AFB) microscopy staining techniques or long turnaround times in gold-standard culture. Therefore, the delays in diagnoses lead to late managements and increased mortalities in TBM, especially in multidrug-resistance (MDR) cases. In the past, a lot of studies tried to solve these problems urgently, but the low frequency of confirmed cases and the absence of a consensus clinical case definition were the huge barriers causing a lack of progression in new clinical trials. In 2010, a uniform clinical case definition for use in clinical research about TBM was established. They used criteria from clinical characteristics, cerebrospinal fluid (CSF) examinations, neuroimaging studies, and evidence of tuberculosis elsewhere. Additionally, microbiological or pathological proof was used to classify the patients who had signs and symptoms of meningitis and were defined as definite, probable, possible, and not tuberculous meningitis. Since then, many clinical studies about TBM diagnosis were developed and made more convenient.

The Xpert MTB/RIF assay was the closed-cartridge-based system heminested PCR for the diagnosis of tuberculosis (TB), and detecting the rifampicin resistant gene in sputum and the CSF. This can be used as a marker for MDR-TB, focused on endemic areas and HIV coinfection. This test has better diagnostic threshold levels (80-100 cfu/ml) than the 5,000 cfu/ml in AFB microscopy staining techniques, shorter duration for the results than conventional TB cultures, and more simplification than nucleic-acid amplification tests. Many studies about the diagnostic accuracy revealed that sensitivity and specificity of this new test varied from 50-86 % and 94-98 % depended on method, population, and laboratory techniques. There were some discussions about the application practicality in the diagnosis of TBM, such as in a large-population study in Vietnam that questioned the lower sensitivity and cost-effectiveness compared with conventional staining and culture. Subsequently, this newer rapid test was approved by WHO for TBM diagnosis.

In Thailand, one of the countries with a high burden of tuberculosis, despite many advantages, use of this test was limited in CSF specimens due to the lack of data, including accuracy in CSF specimens for TBM diagnosis among the Thai population. This study aims to prospectively find out the diagnostic performance and accuracy of Xpert MTB/RIF in CSF samples from patients who presented with subacute lymphocytic meningitis in Northern Thailand, which can be the database for extending the study to cover patients in other parts of Thailand.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of meningitis symptoms and signs including one or more of the following: headache, irritability, vomiting, fever, neck stiff ness, convulsions, focal neurological deficits, altered consciousness, or lethargy at least 5 days prior to admission, plus
2. CSF with abnormalities of at least two of these three characters;

   * Lymphocytic pleocytosis (≥ 50%)
   * More than 40 mg/ml of protein
   * Lower than 0.5 of CSF: blood sugar ratio

Exclusion Criteria:

1. Contraindicated in lumbar puncture
2. Positive for cryptococcal antigen in the CSF.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Detection of M. tuberculosis from CSF specimen | 2 years
  Diagnostic values of Xpert MTB/RIF for detecting M. tuberculosis from CSF

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marais S, Thwaites G, Schoeman JF, Torok ME, Misra UK, Prasad K, Donald PR, Wilkinson RJ, Marais BJ. Tuberculous meningitis: a uniform case definition for use in clinical research. Lancet Infect Dis. 2010 Nov;10(11):803-12. doi: 10.1016/S1473-3099(10)70138-9. Epub 2010 Sep 6. PMID 20822958
- [Background] Marx GE, Chan ED. Tuberculous meningitis: diagnosis and treatment overview. Tuberc Res Treat. 2011;2011:798764. doi: 10.1155/2011/798764. Epub 2011 Dec 21. PMID 22567269
- [Background] Nhu NT, Heemskerk D, Thu do DA, Chau TT, Mai NT, Nghia HD, Loc PP, Ha DT, Merson L, Thinh TT, Day J, Chau Nv, Wolbers M, Farrar J, Caws M. Evaluation of GeneXpert MTB/RIF for diagnosis of tuberculous meningitis. J Clin Microbiol. 2014 Jan;52(1):226-33. doi: 10.1128/JCM.01834-13. Epub 2013 Nov 6. PMID 24197880
- [Background] Patel VB, Theron G, Lenders L, Matinyena B, Connolly C, Singh R, Coovadia Y, Ndung'u T, Dheda K. Diagnostic accuracy of quantitative PCR (Xpert MTB/RIF) for tuberculous meningitis in a high burden setting: a prospective study. PLoS Med. 2013 Oct;10(10):e1001536. doi: 10.1371/journal.pmed.1001536. Epub 2013 Oct 22. PMID 24167451